CLINICAL TRIAL: NCT05232253
Title: Measurement of Bladder Pressure With a Novel External Device (Cystoealstometer) - Home
Brief Title: Cystoealstometer (Bladder Monitor Device)-Home Use
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Christopher Cooper, Associate Dean, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 202010469
Record Dates: First submitted 2022-01-03; First posted 2022-02-09 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Urinary Bladder, Neurogenic
Keywords: urodynamics; neurogenic; bladder
MeSH Terms: conditions — Urinary Bladder, Neurogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Neurogenic Bladder Patient (Experimental): Patients with neurogenic bladder
  Interventions: Device: Cystoelastometer - Urodynamics Testing

INTERVENTIONS:
Device: Cystoelastometer - Urodynamics Testing — The non-invasive cystoelastometer device connects to the drainage end of urinary catheter that the patient uses for routine daily catheterization. Once urine flows into the device a pressure measurement is recorded and stored in the device along with the time and date. The remaining urine is then evacuated through the catheter and device and the cystoelastometer records the volume of urine evacuated. The measurement(s) of bladder pressure and volume as well as the time and date can later be transmitted wirelessly to a smart phone that contains an app for the device.

SUMMARY:
The investigators have developed a novel pressure monitoring device called a 'cystoelastometer' that connects to a drainage end ofastandard urinary catheters that are used by patients with a neurogenic bladder on daily clean intermittent catheterization. The device has already been demonstrated to be accurate in measuring bladder pressure compared to the gold standard urodynamics that are performed in the clinic or hospital. This study will assess the patients and care givers ability and experience using the cystoelastometer device in a home setting.

DETAILED DESCRIPTION:
: For patients with neurogenic bladder, regular monitoring of bladder pressure and capacity is a critical component of maintaining renal and urinary health. This monitoring is currently done by in-office urodynamics testing (UDS). This testing is done intermittently, leaving open the possibility of worsening of bladder function and renal deterioration between testing sessions.

This study utilizes a novel pressure and bladder volume monitoring device which is portable and attaches to the end of a standard urinary catheter and measures the pressure in the device and then assists in the drainage of the bladder and records the bladder volume. The investigators will be investigating if this device can be used by patients or their caregivers in a home setting.

This study will enroll patients with neurogenic bladder that currently perform clean intermittent catheterization on a daily basis as part of their regular care. The patients will be asked to use the device at least twice a day for two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients seen in the University of Iowa Pediatric Urology Clinic with neurogenic bladder managed with clean intermittent catheterization.
* Patients who haven't had any change in management
* Patients who had recently had UDS (urodynamic study) performed

Exclusion Criteria:

* phone which is not iOS compatible

Ages: 6 Months to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Home use of bladder pressure and volume monitoring device- Cystoelastometer | Two weeks
  Utilization study of novel external cystoelastometer device - Home bladder pressure and volume monitor recorded in terms of cm H2O pressure and urine evacuation device with volume measurement in terms of milliliters.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher S Cooper, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospital and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No